Efficacy of Ulipristal Acetate in Induction of Second Trimestric Missed Abortion in Women with Previous Caesarian section: Randomized Controlled Trial.

**Document date: February 2020** 

## Statistical analysis:

The collected data were coded, tabulated, and statistically analyzed using IBM SPSS statistics (Statistical Package for Social Sciences) software version 22.0, IBM Corp., Chicago, USA, 2013. Quantitative normally distributed data described as mean±SD (standard deviation) after testing for normality using Shapiro-Wilk test, then compared using independent t-test if normally distributed and Mann Whitney test if not normally distributed, while Pearson test was used for correlations. Qualitative data described as number and percentage and compared using Chi square test and Fisher's Exact test for variables with small expected numbers. Log rank test was used to compare abortion rate. The level of significance was taken at P value < 0.050 was significant, otherwise was non-significant